CLINICAL TRIAL: NCT00504764
Title: APL-R2007: Treatment of Relapsed Promyelocytic Leukemia With Arsenic Trioxide (ATO)
Brief Title: Treatment of Relapsed Promyelocytic Leukemia With Arsenic Trioxide (ATO)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAP-R2007
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Relapsed Acute Promyelocytic Leukemia; Arsenic Trioxide
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide; Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Arsenic Trioxide — Induction ATO 0.15 mg/kg/day IV until CR or a maximum of 60 days In isolated molecular relapse ATO will be administered at same dose, 5 days a week, during 6 weeks.
  Consolidation ATO 0.15 mg/kg/day IV 5 days week, during 5 weeks
Procedure: Autologous Transplantation — Autologous Transplantation
Procedure: Allogenic Transplantation — Allogenic Transplantation
Drug: ATRA — Consolidation: ATRA 45 mg/m²/day oral during 5 weeks

SUMMARY:
Summary Acute promyelocytic leukemia is defined by a characteristic morphology (AML FAB M3/M3v), by the specific translocation t(15;17) and its molecular correlates (PML/RARa and RARa/PML). Thereby it can be separated from all other forms of acute leukemia.

By all-trans retinoic acid in combination with chemotherapy cure rates of 70 to 80% can be reached. On average, about 10% of patients still die in the early phase of the treatment and about 20 to 30% relapse. Molecular monitoring of the minimal residual disease (MRD) by qualitative nested RT-PCR and quantitative REAL-time PCR of PML/RARa allows to follow the individual kinetics of MRD and to identify patients with an imminent hematological relapse.

A standardized treatment for patients with relapsed APL has not yet been established. With arsenic trioxide (ATO) monotherapy remission rates over 80% were achieved and long-lasting molecular remissions are described. The drug was mostly well tolerated. ATO exerts a dose dependent dual effect on APL blasts, apoptosis in higher and partial differentiation in lower concentrations. ATO was also successfully administered before allogeneic and autologous transplantation. ATO is approved for the treatment of relapsed and refractory APL in Europe and in the USA.

After remission induction, there are several options for postremission therapy Previous studies shows that risk of relapse is higher in patients treated with ATO postremission in monotherapy , than in other that receive ATO plus chemotherapy or transplantation (TPH). Also, compared with chemotherapy, ATO induction and consolidation has a favorable impact in posterior response to transplantation. It is due to a low toxicity or a best quality of remission to TPH. It seems better, for these reasons, the intensification with TPH (autologous or allogenic) in patients with relapsed APL treated with ATO. For another hand, patients no candidates to TPH can be treated with ATO combined with other active agents in APL, as ATRA, anthracyclines o Mylotarg

DETAILED DESCRIPTION:
Induction ATO 0.15 mg/kg/día IV in continuous perfusion 1-2 hours/day until complete response (CR) or maximum of 60 days.

Oral hydroxyurea treatment (initial dose 2 g/day)is recommended in patients with leucocyte counts at relapse >10x109/L or in the two first weeks of induction.

Isolated molecular relapsed patients will be treated with ATO (same dose) 5 days at week, during 6 weeks.

Consolidation ATO 0.15 mg/kg/día IV 5 days at week, during 5 weeks, combined with oral ATRA 45 mg/m²/day during the same 5 weeks.

Post-consolidation therapy TPH (autologous or allogenic) in candidate patients. In case of molecular remission, is recommended autologous-TPH.

Patients no candidates to auto-TPH or alo-TPH, should will follow treatment with ATO cycles + ATRA +/- Mylotarg.

1. Option Alo-TPH If PCR post-consolidation is negative is recommended auto-TPH. However, if alo-TPH is decided, it will be done immediately without preceding chemotherapy.

   If PCR post-consolidation is positive, should done alo-TPH.
2. Option Auto-TPH If PCR post-consolidation is negative it will be administered one cycle of MTZ + Ara-C follow by auto-TPH.

   In cas of failure: a) if patient has autologous stem cells preserved (PCR negative) are suitable for auto-TPH; b) patients with HLA-compatible donor who are suitable for allogenic stem cell transplantation should be transplanted; c) Patients who are not eligible for allogenic or autologous transplantation, receive various cycles with ATO + ATRA combined or not with Mylotarg.

   If PCR post-consolidation is positive and patient is eligible for allogenic TPH, should be done a allogenic TPH.

   If patient is no eligible for allogenic TPH or dont has compatible donor, will be administrate one cycle of MTZ + Ara-C and collect stem cells. Autologous transplantation will be done if after this cycle, a molecular remission is obtained. No molecular remission or no enough stem cells collection, patient follows treatment with subsequent cycles of ATO + ATRA combined or no with Mylotarg.
3. ATO + ATRA combined or no with Mylotarg Patients no eligible to autologous TPH or allogenic TPH follows treatment with subsequent cycles of ATO + ATRA combined or no with Mylotarg.

If Mylotarg is no possible, treatment will be with subsequent cycles of ATO + ATRA.

ATO + ATRA + Mylotarg: Mylotarg 6 mg/m2 day 1, ATO 0.15 mg/kg days 1 to 5 and 8 to 12, and ATRA 45 mg/m2/d days 1 to 15. Doses of mylotarg should be reduced to 3 mg/m2 in patients aged over 60 years. Administration of 3 cycles with a month interval, follow of 3 to 6 cycles of ATO + ATRA without Mylotarg. After, ATRA 45 mg/m2/d 15 days every 3 months until complete two years of maintenance.

ATO + ATRA: ATO 0.15 mg/kg days 1 to 5 and 8 to 12, and ATRA 45 mg/m2/d days 1 to 15, every 29 days. Administration of 9 cycles, and followed by ATRA 45 mg/m2/d during 15 days every 3 months until complete two years of maintenance.

ELIGIBILITY:
Inclusion Criteria:

* ECOG ≤ 3.
* Patients in first or subsequent hematological or molecular relapse of APL
* Persistence of a positive PCR (positive PCR after 3 consolidation cycles of first line therapy).
* Diagnostic measures Confirmation of relapse by RT-PCR of PML/RARa, cytogenetics, FISH or positive PGM3.
* Age over 18 years (No upper age limit)
* Informed consent of the patient

Exclusion Criteria:

* ECOG 4.
* Heart failure NYHA grade III and IV.
* Renal or hepatic failure WHO grade ³III
* Positive HIV.
* Psychological dysfunction
* Associated active neoplasia
* Pregnancy.
* Arsenic Hypersensibility.
* QTc-interval prolonged over 460 msec before therapy (normal electrolytes, no other drugs prolonging the QT-interval )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the hematological and molecular remission rate after induction and consolidation with ATO | 1 year
Evaluate the induction mortality with ATO in monotherapy | 1 year
Evaluate the hematological and molecular relapse rate in patients treated with autologous transplantation, allogenic transplantation or ATO + ATRA +/- Mylotarg | 1 year

SECONDARY OUTCOMES:
Evaluate kinetics of the MDR of PML/RARa during and after ATO | 2 years
Evaluate the mortality related with postremission treatment | 1 year
Side effects of ATO and the different treatments post-consolidation | 2 years
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sanz Miguel Angel, Dr, Study Chair — Hospital La Fe; Esteve Jordi, Dr, Study Chair — Hospital Clinic of Barcelona; Montesinos Pau, Dr, Study Chair — Hospital General Universitario de Valencia
Locations (86):
- Spain (86):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital Ntra. Sra. Sonsoles, Ávila, Avila
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Valle Hebrón, Barcelona, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital general de Castellón, Castelló, Castellón
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Complejo Hospitalario Reina Sofía, Córdoba, Córdoba
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hospital Médico Quirúrgico Ciudad de Jaén, Jaén, Jaen
  - Hospital Juan Canalejo, A Coruña, La Coruña
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital Arnau de Vilanova, Lleida, Lleida
  - Hospital de Alcorcón, Alcorcón, Madrid
  - Clínica La Concepción, Madrid, Madrid
  - Clínica Puerta de Hierro, Madrid, Madrid
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid, Madrid
  - . Hospital Clínico Universitario Virgen de la Victoria, Málaga, Málaga
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital del Río Carrión, Palencia, Palencia
  - Hospital Son Dureta, Palma de Mallorca, Palma de Mallorca
  - Hospital Son Llàtzer, Palma de Mallorca, Palma de Mallorca
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Joan XXIII, Tarragona, Tarragona
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Hospital Clínic, Valencia, Valencia
  - Hospital General Universitario, Valencia, Valencia
  - Hospital La Fe, Valencia, Valencia
  - Complejo Hospitalario Xeral-Cies, Vigo, Vigo
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Fundación Hospital Alcorcón, Alcorcón
  - Hospital de la Ribera, Alzira
  - Hospital Clinic, Barcelona
  - Basurtuko Ospitalea, Basurto
  - Hospital de Cruces, Bilbao
  - Complejo Hospitalario de Cáceres, Cáceres
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital General de Elda, Elda
  - Hospital de Fuenlabrada, Fuenlabrada
  - Hospital General de Guadalajara, Guadalajara
  - Area Hospitalaria Juan Ramón Jimenez, Huelva
  - Hospital de San Jorge, Huesca
  - Hospital de Jerez de la Frontera, Jerez de la Frontera
  - Hospital General de Lanzarote, Lanzarote
  - Complejo Hospitalario León, León
  - Complexo Hospitalario Xeral-Calde, Lugo
  - Clínica Moncloa, Madrid
  - Clínica Puerta de Hierro, Madrid
  - Clínica Rúber, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Central de la Defensa, Madrid
  - Hospital de la Princesa, Madrid
  - Hospital Doce de Octubre, Madrid
  - Hospital la Paz, Madrid
  - Althaia, Xarxa Asistencial de Manresa, Manresa
  - Fundación Hospital Sant Joan de Déu de Martorell, Martorell
  - Hospital de Mérida, Mérida
  - Hospital de Móstoles, Móstoles
  - Hospital General Morales Meseguer, Murcia
  - Hospital de Gran Canaria Doctor Negrín, Palma de Gran Canaria
  - Hospital Verge del Toro, Palma de Mallorca
  - Complejo Hospitalario de Pontevedra_Hospital Montecelo, Pontevedra
  - Complejo Hospitalario de Pontevedra_Hospital Provincial, Pontevedra
  - Corporació Sanitaria Parc Taulí, Sabadell
  - Hospital de Sagunto, Sagunto
  - Hospital Clínico de Salamanca, Salamanca
  - Clínica Sant Camil, Sant Pere de Ribes
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital General de Segovia, Segovia
  - H.U. Virgen del Rocio, Seville
  - Hospital Nuestra Señora del Prado, Toledo
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Dr. Peset, Valencia
  - Hospital Francesc de Borja, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Hospital Comarcal Pius de Valls, Valls
  - Comarcal de Vinaros, Vinaròs
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital de Galdakao, Vizcaya
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- See also: Spanish association of Haematology — http://www.aehh.org